CLINICAL TRIAL: NCT00545857
Title: Effect of Pioglitazone on the Course of New Onset Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Thomas A. Wilson, Professor of Pediatrics, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20064114
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes; Insulin dependent diabetes; Juvenile onset diabetes; pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: pioglitazone; Drug: Placebo control
- Placebo control (Placebo Comparator)
  Interventions: Drug: pioglitazone; Drug: Placebo control

INTERVENTIONS:
Drug: pioglitazone — Pioglitazone daily; dose varies with size
  Other Names: Actos
Drug: Placebo control — Comparison of pioglitazone vs. placebo on the outcome of type 1 diabetes mellitus
  Other Names: Actos

SUMMARY:
A study to examine the effect of pioglitazone on the course of new onset type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Thiazolidinediones have been shown to reduce the development of diabetes mellitus in animal models of type 1 diabetes and to reduce the death of beta cells (cells that make insulin) in petri dishes. Pioglitazone is a thiazolidinedione currently approved for the treatment of type 2 diabetes. This study explores the question of whether pioglitazone can preserve beta cell function in patients with recently diagnosed type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes mellitus diagnosed within 4 months
* Age > 6 years of age
* Ability to swallow capsule
* Signed informed consent / assent

Exclusion Criteria:

* Other illnesses

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2002-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
C-peptide response to a Sustacal meal | 6 months

SECONDARY OUTCOMES:
Insulin requirement | 6 months
Hemoglobin A1c | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Wilson, MD, Principal Investigator — State University of New York Stony Brook
Locations (1):
- Thomas A. Wilson, MD, Stony Brook, New York, United States

REFERENCES:
- [Derived] Tafuri KS, Godil MA, Lane AH, Wilson TA. Effect of pioglitazone on the course of new-onset type 1 diabetes mellitus. J Clin Res Pediatr Endocrinol. 2013;5(4):236-9. doi: 10.4274/Jcrpe.981. PMID 24379032